CLINICAL TRIAL: NCT00736164
Title: A Randomized, Double Blind, Placebo Controlled Clinical Trial of Supplementation of L-Selenomethionine in Patients With Prostate Cancer Prior to Prostatectomy or Brachytherapy (Se Pre-Prostatectomy/Pre-Brachytherapy Trial)
Brief Title: Selenomethionine in Treating Patients Undergoing Surgery or Internal Radiation Therapy for Stage I or Stage II Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No accrual
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: James L. Mohler, Roswell Park Cancer Institute
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000611981; P30CA016056 (NIH); RPCI-I-104307
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2012-02-06 (Estimated); Status verified 2012-02

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage II prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Selenomethionine

ARMS (2):
- Arm I (Experimental): Patients receive oral selenomethionine once daily for 8-9 weeks.
  Interventions: Dietary Supplement: selenomethionine
- Arm II (Placebo Comparator): Patients receive oral placebo once daily for 8-9 weeks.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: selenomethionine — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Selenomethionine may slow the growth of prostate cancer. Giving selenomethionine before surgery or internal radiation therapy may be an effective treatment for prostate cancer.

PURPOSE: This randomized phase II trial is studying how well selenomethionine works in treating patients undergoing surgery or internal radiation therapy for stage I or stage II prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To investigate the down-regulation of the androgen receptor using tissue samples from patients with stage I or II prostate cancer treated with selenomethionine for 8-9 weeks prior to undergoing prostatectomy or brachytherapy.

Secondary

* To evaluate the down regulation of a number of genes regulated by the androgen receptor (i.e., prostate-specific antigen, kallikrein 2, cell division cycle 6, and dehydrocholesterol reductase 24) using tissue samples from these patients.
* To evaluate the down-regulation of haptic nuclear factor 3-alpha using tissue samples from these patients.
* To evaluate whether the thiol methyltransferase phenotype modifies the prostatic response to short-term selenomethionine supplementation in these patients.

Tertiary

* To use quantitative nuclear morphometry to index cellular abnormality in tissue samples as measured by nuclear texture (e.g., total optical density, nuclear area, mean nuclear density, and optical heterogeneity).

OUTLINE: Patients are stratified according to planned treatment (brachytherapy vs prostatectomy). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral selenomethionine once daily for 8-9 weeks. Patients then undergo prostatectomy or brachytherapy.
* Arm II: Patients receive oral placebo once daily for 8-9 weeks. Patients then undergo prostatectomy or brachytherapy.

Blood samples are collected at baseline and on the day of prostatectomy or brachytherapy. Samples are analyzed for selenium accumulation by atomic absorption spectrophotometry. Additional blood samples are stored for future analysis of alpha tocopherol, lycopene, and other vitamin levels, as well as oxidative stress biomarkers. Selenium accumulation is also evaluated in toenail samples at baseline to assess long-term selenium status. Prostate tissue samples are obtained during prostatectomy or brachytherapy and analyzed for RNA and expression of selenium-linked biomarkers (e.g., androgen receptor, prostate-specific antigen, kallikrein 2, cell division cycle 6, dehydrocholesterol reductase 24, and haptic nuclear factor 3 alpha) by quantitative reverse transcription (RT)-PCR. Biomarker expression is compared in both prostatectomy and brachytherapy specimens.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Diagnosed by sextant or greater biopsy
  * Clinical stage T1a-T2c disease
* Gleason score < 8
* Prostate-specific antigen < 20.0 ng/mL
* Scheduled to undergo prostatectomy or brachytherapy

PATIENT CHARACTERISTICS:

* Life expectancy > 5 years
* No other prior malignancy except nonmelanoma skin cancer
* Willing to take selenomethionine or placebo for 8-9 weeks immediately prior to undergoing prostatectomy or brachytherapy

PRIOR CONCURRENT THERAPY:

* No prior hormonal therapy or radiotherapy
* More than 30 days since prior and no concurrent participation in any other clinical trial involving a medical, surgical, nutritional, or lifestyle intervention (e.g., dietary modification or exercise)
* No concurrent dietary supplementation with selenium at doses > 60 mcg/day, including multivitamin supplements
* No concurrent hormonal therapy, including 5-alpha reductase inhibitors (e.g., finasteride or dutasteride); anti-androgens (e.g., bicalutamide, flutamide, or ketoconazole); or luteinizing hormone-releasing hormone agonists (e.g., leuprolide acetate, goserelin acetate, or abarelix)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Quantity of androgen receptor message expression

SECONDARY OUTCOMES:
Expression of prostate-specific antigen, kallikrein 2, cell division cycle 6, and dehydrocholesterol reductase 24
Expression of haptic nuclear factor 3-alpha
Variation in thiol methyltransferase phenotype

CONTACTS AND LOCATIONS:
Overall Officials: James L. Mohler, MD, Principal Investigator — Roswell Park Cancer Institute